CLINICAL TRIAL: NCT06911333
Title: A Phase I/IIa Trial of AD1208, a Cell Cycle Inhibitor/MASTL Inhibitor, as a Single Agent or a Combination in Subjects With Any Progressive, Locally Advanced(Unresectable) or Metastatic Solid Tumors
Brief Title: AD1208 in Subjects With Any Progressive, Locally Advanced or Metastatic Solid Tumors
Acronym: AD1208
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avelos Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AVS1001-101
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult; Tumor, Solid; Solid Tumor; Solid Tumor, Unspecified, Adult; Solid Tumor Cancer; Solid Tumors Refractory to Standard Therapy; Solid Tumor in Advanced Stage
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 (Experimental): AD1208 dose 1 (40mg bid) treatment arm
  Interventions: Drug: AD1208
- Cohort 2 (Experimental): AD1208 dose 2 (80mg QD) treatment arm
  Interventions: Drug: AD1208
- Cohort 3 (Experimental): AD1208 dose 3 (80mg bid) treatment arm
  Interventions: Drug: AD1208
- Cohort 4 (Experimental): AD1208 dose 4 (140mg bid) treatment arm
  Interventions: Drug: AD1208
- Cohort 5 (Experimental): AD1208 dose 5 (240mg bid) treatment arm
  Interventions: Drug: AD1208
- Cohort 6 (Experimental): AD1208 dose 6 (340mg bid) treatment arm
  Interventions: Drug: AD1208

INTERVENTIONS:
Drug: AD1208 — Up to 6 of cohorts will be applied sequentially in phase Ia part.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and tolerability of AD1208 to determine the maximum tolerated dose(MTD) or maximumly administered dose(MAD) in any progressive, locally advanced (unresectable) or metastatic solid tumors. The main questions it aims to answer are:

* Which dosage of AD1208 is safe and tolerable for participants?
* What medical problems do participants have when taking AD1208?

Participants will:

* Take drug AD1208 every day up to 1 cycle at the least.
* Visit the site once every 1 weeks for checkups and tests during cycle 1 and every 3 weeks from cycle 2 onwards.
* Keep a diary of any adverse events and administrated drug

DETAILED DESCRIPTION:
- Dose-escalation Part The treatment cycle is defined as 21 days and AD1208 will be administered orally once or twice a day from Day 1 to Day 21 in every 21-day cycle. The dose-escalation part is divided into phase 1a, which determines the Recommended dose of AD1208 in monotherapy, and phase 1b, which determines the RP2D of AD1208 in combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects ≥19 years of age
* Willing to consent to participate in study and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures
* Histologically and/or cytologically confirmed any progressive, locally advanced (unresectable), or metastatic solid tumors that have relapsed or are refractory following the last line of treatment and for which prior standard therapy has been ineffective, standard therapy does not exist or is not considered appropriate.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Life expectancy of at least 12 weeks
* Subjects with adequate hematologic, hepatic, and renal functions confirmed based on the screening laboratory test within 2 weeks prior to the first administration of IP.
* Female subject who is surgically sterile, is postmenopausal, or agrees to use a highly effective method of birth control (2 methods strongly recommended) during the study and for 6 months following the last dose of IP.
* Male subject with a pregnant or breastfeeding partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy or for the time the partner is breastfeeding throughout the study period and for 6 months after the final administration of IP.

Exclusion Criteria:

* Untreated active brain metastases.
* has leptomeningeal disease.
* unrecovered > Grade 1 from the adverse event of prior therapy except for alopecia.
* has an active autoimmune disease requiring systemic treatment within the past 2 years.
* Active interstitial lung disease (ILD) or pneumonitis or a history of ILD.
* Subject has received the following treatment;

  * prior anticancer monoclonal antibody treatment or investigational therapy
  * prior any chemotherapy
  * prior radiotherapy
  * Major surgery
* Clinically significant (i.e., active) cardiovascular disease
* known positive of human immunodeficiency virus (HIV) infection.
* Active hepatitis B or C subjects.
* known allergic reaction for active ingredients or inactive ingredients such as excipients of Investigational product.
* Live vaccine administered against infectious disease.
* Gastrointestinal (GI) track disease causing the inability to take oral medication, malabsorption syndrome or uncontrolled inflammatory GI disease.
* having psychiatric illness/social situations that would limit compliance with study requirements.
* women with a positive pregnancy test at screening test.
* women who are breast feeding.
* subject has any condition because of which, in the opinion of the investigator, the participation would not be in the best interest of the subject.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2030-02-20 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | At the end of Cycle 1 (each cycle is 21 days)
  to determine maximum tolerated dose (MTD) or maximumly administered dose (MAD)

SECONDARY OUTCOMES:
Maximum Plasma Concentration [Cmax] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
A trough level or trough concentration [Ctrough] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
Time to peak drug concentration [Tmax] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
Half-life [T1/2] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
The area under the curve up to the last quantifiable time-point [AUC0-last] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
Clearance [CL] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
Volume of distribution at steady state [Vss] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to characterize pharmacokinetic profile of AD1208
objective response rate [ORR] | through study completion, an average of 1 year
  to evaluate the preliminary antitumor activity
disease control rate [DCR] | through study completion, an average of 1 year
  to evaluate the preliminary antitumor activity
treatment duration | through study completion, an average of 1 year
  to evaluate the preliminary antitumor activity
progression-free survival [PFS] | through study completion, an average of 1 year
  to evaluate the preliminary antitumor activity

OTHER OUTCOMES:
metabolite 6 [M6] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to profile the metabolites of AD1208
metabolite 8 [M8] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to profile the metabolites of AD1208
metabolite 9 [M9] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to profile the metabolites of AD1208
metabolite 10 [M10] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to profile the metabolites of AD1208
metabolite 11 [M11] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to profile the metabolites of AD1208
metabolite 12 [M12] | At the Day 1 and Day 15 of Cycle 1 (each cycle is 21 days)
  to profile the metabolites of AD1208
PPP2R2A | baseline, pre-intervention/procedure/surgery
  to investigate Potential predictive biomarker related to AD1208

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Severance Hospital, Seoul
  - Samsung Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No